CLINICAL TRIAL: NCT02501655
Title: ANALYSIS OF DEPOSITION RADIOAEROSOL NEBULIZERS MEMBRANE IN HEALTHY SUBJECTS
Brief Title: Analysis of Deposition With Nebulizers Membrane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daniella Cunha Brandao (Other)
Responsible Party: Sponsor-Investigator, Daniella Cunha Brandao, Daniella Cunha Brandão, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Luciana doutorado 01
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1 (Active Comparator): Jet Nebulizer - control group
  Interventions: Device: Phase 2- mesh nebulizer
- Phase 2 (Experimental): Mesh nebulizers
  Interventions: Device: phase 1 - jet nebulizer

INTERVENTIONS:
Device: phase 1 - jet nebulizer — Aerosol generators diethilene penta-acetic triamine technetium (99mTc-DTPA) with radioactivity of 1 millicuries (Noble et al., 2007) mixed with 0.9% saline solution with a total volume of 4 ml using jet nebulizer (NS - mark) and 8l/min of the oxygen
  Arms: Phase 2
Device: Phase 2- mesh nebulizer — Aerosol generators diethilene penta-acetic triamine technetium (99mTc-DTPA) with radioactivity of 1 millicuries (Noble et al., 2007) mixed with 0.9% saline solution with a total volume of 2 ml using vibrating mesh inhaler with valved chamber adapter (Aerogen Solo with Ultra Adapter, Aerogen Ltd).
  Arms: Phase 1

SUMMARY:
BACKGROUND: Mesh nebulizers (MN) have lower residual volume and increased inhaled dose compared to jet nebulizers (JN) per in vitro and animal models. The aim of this study was to compare radioaerosol deposition using MN and JN in healthy subjects, using 2-D planar scintigraphy. METHODS: A randomized trial in 6 normal subjects (4 female, 2 male) inhaled 99mTc-DTPA with an activity of 1 mCi with the normal saline to a total dose of 4 mL with JN (Misty Max, Air Life, Yorba Linda, USA) oxygen flow of 8 L / min and 1.5 mL with MN (Aeroneb Solo with Ultra adapter; Aerogen Galway, Ireland). Scintigraphy was used to determine distribution of deposition and mass balance between compartments.

ELIGIBILITY:
Inclusion Criteria:

* The study inclusion critera was healthy adults of both sexes, between 18 to 65 years, without history of lung disease or smoking, with forced vital capacity (FVC) or forced expiratory volume in the first second (FEV1) greater or equal to 80% of predicted values (Pereira et al., 1992), ability to follow and retain verbal commands while able and willing to provide signed consent to participate in this study.

Exclusion Criteria:

* Participants were excluded if they have been diagnosed with a lung disease, current smoker, unable to understand and follow the procedures and pregnant or unable to tolerate nebulization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
radioaerosol deposition index into the lungs | 1 month
  Immediately after inhalation, participants sat in a chair with the back positioned in front to the gamma camera (STARCAM 3200 GE, California, USA) to obtain radioactivity counts from the posterior thorax during a period of 300 seconds on a matrix of 256 X 256. After, participants were positioned sitting in front to the gama camera to obtain images from face. Then, the same procedure was performed to analysis deposition in the nebulizer, circuits, inspiratory filter, expiratory filter and face mask. Counts representing stomach were obtained from posterior thorax and corrections for decay of technetium were used to during extrapulmonary measurements

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Alcoforado, Principal Investigator — UFPE
Locations (1):
- Hospital das Clínicas de Pernambuco, Recife, Pernambuco, Brazil